CLINICAL TRIAL: NCT01265433
Title: Randomized Phase II Study of Adjuvant WT-1 Analog Peptide Vaccine in Patients With Malignant Pleural Mesothelioma (MPM) After Completion of Combined Modality Therapy
Brief Title: Galinpepimut-S (WT-1 Analog Peptide) Vaccine in Malignant Pleural Mesothelioma After Combined Modality Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sellas Life Sciences Group (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-134; NCT01890980 (obsolete NCT alias)
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: GM-CSF; MONTANIDE ISA 51; WT1 PEPTIDE SPECIFIC T CELLS; Vaccine; 10-134; Galinpepimut-S
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Monatide (IMS 3015); Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galinpepimut-S + Montanide + GM-CSF (Experimental): Galinpepimut-S emulsified with Montanide adjuvant (1:1 ratio) 1 mL and GM-CSF 70 mcg
  Interventions: Biological: Galinpepimut-S + Montanide + GM-CSF
- Montanide + GM-CSF (Placebo Comparator): Montanide adjuvant 1 mL and GM-CSF 70 mcg
  Interventions: Biological: Montanide + GM-CSF

INTERVENTIONS:
Biological: Galinpepimut-S + Montanide + GM-CSF — Patients will receive 6 injections over 12 weeks. Treatment will be administered on weeks 0, 2, 4, 6, 8, and 10. All patients will receive Sargramostim (GM-CSF) (70 mcg) injected subcutaneously on days 0 and -2 of each vaccination. Patients may self administer the Sargramostim (GM-CSF) on day -2 if they have been appropriately instructed on SQ injection administration. Patients will be informed of the expected reactions such as irritation at the injection site. Patients will keep a logbook noting the time and placement of the injection. Patients will also receive 1.0 ml of emulsion with Montanide alone or with WT-1 peptides plus Montanide. It will be administered by a nurse (it may not be self administered) subcutaneously to the same anatomical site as the GM-CSF. This site will be marked by the patient or treating healthcare professional by a permanent marker pen.
  Arms: Galinpepimut-S + Montanide + GM-CSF
Biological: Montanide + GM-CSF — Patients will receive 6 injections over 12 weeks. Treatment will be administered on weeks 0, 2, 4, 6, 8, and 10. All patients will receive Sargramostim (GM-CSF) (70 mcg) injected subcutaneously on days 0 and -2 of each vaccination. Patients may self administer the Sargramostim (GM-CSF) on day -2 if they have been appropriately instructed on SQ injection administration. Patients will be informed of the expected reactions such as irritation at the injection site. Patients will keep a logbook noting the time and placement of the injection. Patients will also receive 1.0 ml of emulsion with Montanide alone or with WT-1 peptides plus Montanide. It will be administered by a nurse (it may not be self-administered)subcutaneously to the same anatomical site as the GM-CSF. This site will be marked by the patient or treating healthcare professional by a permanent marker pen.
  Arms: Montanide + GM-CSF

SUMMARY:
Study of galinpepimut-S, a Wilms Tumor-1 (WT1) vaccine, to see if it delays or prevents the mesothelioma from growing back after surgery. WT1 is a protein in cancer cells that regulates gene expression and causes cell growth.

DETAILED DESCRIPTION:
The doctors are testing galinpepimut-S, a Wilms Tumor-1 (WT1) vaccine, to see if it delays or prevents the mesothelioma from growing back after surgery. WT1 is a protein in cancer cells that regulates gene expression and causes cell growth. Mesothelioma tumors generally have high levels of WT1.This study was originally designed to have two treatment groups. One group received non-specific immunotherapy with medications called Montanide and Sargramostim (Granulocyte Macrophage Colony Stimulating Factor, GM-CSF). Enrollment to this group has stopped The other group, which continues receives more specific immunotherapy with galinpepimut-S plus Montanide and GM-CSF. Both Montanide and GM-CSF are commonly given along with vaccines because they have a general effect in boosting the immune response. Some researchers believe that this general increase in the immune system may have some effect in treating cancer. Some studies using GM-CSF with melanoma vaccines have suggested that it could lessen the effects of the vaccine. The addition of the WT1 proteins makes this therapy more directed to mesothelioma. The combination of galinpepimut-S with Montanide and GM-CSF has been tested in a prior trial including 9 patients with advanced mesothelioma. In that trial, the vaccine was safe and caused an immune response.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of malignant pleural mesothelioma (MPM) confirmed at participating institution.
* Positive immunohistochemical staining for WT-1 (greater than 10% of cells).
* Completion of multimodality therapy. This must include surgical resection by either pleurectomy/decortication or extrapleural pneumonectomy. The surgery should be performed with the intent of complete resection, though patients with an R1 resection will still be eligible. Patients should have also received treatment with chemotherapy and/or radiation. Patients with an R2 resection are also eligible as long as the site of residual disease is treated post-operatively with radiotherapy.
* 4-12 weeks since completion of combined modality therapy.
* Age > or = to 18 years
* Karnofsky performance status > or = to 70%
* Hematologic parameters: Absolute neutrophil count > or = to 1000/mcL, Platelets > or = to 50K/mcL.
* Biochemical parameters: Total bilirubin < or = to 2.0 mg/dl, AST and ALT < or = to 2.5 x upper limits of normal, Creatinine < or = to 2.0 mg/dl.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with active infection requiring systemic antibiotics, antiviral, or antifungal treatments.
* Patients with a serious unstable medical illness or another active cancer.
* Patients taking systemic corticosteroids.
* Patients with an immunodeficiency syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-12-21 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Zauderer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zauderer MG, Tsao AS, Dao T, Panageas K, Lai WV, Rimner A, Rusch VW, Adusumilli PS, Ginsberg MS, Gomez D, Rice D, Mehran R, Scheinberg DA, Krug LM. A Randomized Phase II Trial of Adjuvant Galinpepimut-S, WT-1 Analogue Peptide Vaccine, After Multimodality Therapy for Patients with Malignant Pleural Mesothelioma. Clin Cancer Res. 2017 Dec 15;23(24):7483-7489. doi: 10.1158/1078-0432.CCR-17-2169. Epub 2017 Sep 28. PMID 28972039
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Montanide + GM-CSF: Montanide adjuvant + GM-CSF: Patients will receive 6 injections over 12 weeks. Treatment will be administered on weeks 0, 2, 4, 6, 8, and 10. All patients will receive Sargramostim (GM-CSF) (70 mcg) injected subcutaneously on days 0 and -2 of each vaccination. Patients may self administer the Sargramostim (GM-CSF) on day -2 if they have been appropriately instructed on SQ injection administration. Patients will be informed of the expected reactions such as irritation at the injection site. Patients will keep a logbook noting the time and placement of the injection. Patients will also receive 1.0 ml of emulsion with Montanide alone or with WT-1 peptides plus Montanide. It will be administered by a nurse (it may not be self-administered)subcutaneously to the same anatomical site as the GM-CSF. This site will be marked by the patient or treating healthcare professional by a permanent marker pen.
Period: Overall Study
Arm/Group | Galinpepimut-S + Montanide + GM-CSF | Montanide + GM-CSF
Started | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Galinpepimut-S: Galinpepimut-s + Montanide + GM-CSF
- Control: Montanide + GM-CSF
- Total: Total of all reporting groups
Arm/Group | Galinpepimut-S | Control | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Median (Full Range); unit: years] | 70 [34 to 84] | 67 [48 to 79] | 68 [34 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 17 | 18 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Karnofsky performance status at enrollment [Count of Participants; unit: Participants] — The Karnofsky Performance Scale Index classifies the patient's functional impairment, used to assess the prognosis in individual patients. The lower the score, the worse the prognosis.
  100: Able to carry on normal activity; no special care needed. No evidence of disease 90: Able to carry on normal activity; minor signs/symptoms of disease 80: Normal activity with effort; some signs/symptoms of disease 70: Cares for self; unable to carry on normal activity 60: Requires occasional assistance, but able to care of personal needs 50: Requires considerable assistance and frequent medical care
  Participants
    70% | 1 | 3 | 4
    80% | 7 | 12 | 19
    90% | 11 | 6 | 17
    100% | 1 | 0 | 1
Smoking status [Count of Participants; unit: Participants]
  Former | 12 | 13 | 25
  Current | 0 | 0 | 0
  Never | 8 | 8 | 16
Histology [Count of Participants; unit: Participants]
  Epithelioid | 18 | 21 | 39
  Mixed | 2 | 0 | 2
  Sarcomatoid | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 1-year Progression-free Survival
Description: Progression free survival (PFS) rate will be calculated from the time of randomization to first evidence of disease recurrence or death of any cause.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Galinpepimut-S | Control
Number analyzed (Participants) | 20 | 21
percentage of participants | 44 | 33

2. Primary Outcome: Progression-free Survival
Description: Median progression free survival (PFS) is where PFS are assessed from the time of randomization to first evidence of disease recurrence or death of any cause.
Time Frame: Up to 5 years and 11 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Galinpepimut-S | Control
Number analyzed (Participants) | 20 | 21
months | 10.1 [5.5 to 20.8] | 7.4 [2.8 to 14.6]

3. Secondary Outcome: Overall Survival
Description: Median overall survival (OS) is estimated from time of randomization to all cause mortality
Time Frame: Uo to 5 years and 11 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Galinpepimut-S | Control
Number analyzed (Participants) | 20 | 21
months | 22.8 [9.1 to 37.6] | 18.3 [10.2 to 28]

4. Secondary Outcome: Immune Response
Description: Immunogenicity of galinpepimut-S and control from a subset of participants
Time Frame: 12 weeks
Population: Data were available from 22 participants only
Measure: Count of Participants; unit: Participants
Arm/Group | Galinpepimut-S | Control
Number analyzed (Participants) | 10 | 12
Participants
  CD4 Elispot: Positive | 4 | 1
  CD4 Elispot: Negative | 4 | 8
  CD4 Elispot: Not tested | 2 | 3
  CD8 Elispot: Positive | 1 | 1
  CD8 Elispot: Negative | 1 | 3
  CD8 Elispot: Not tested | 8 | 8
  Tetramer assay positive: Positive | 1 | 2
  Tetramer assay positive: Negative | 0 | 3
  Tetramer assay positive: Not tested | 9 | 7

ADVERSE EVENTS:
Time Frame: Up to 5 years and 11 months, from either start of study or randomization, until primary completion (Nov 2016)
Arm/Group | Galinpepimut-S | Control
All-Cause Mortality (participants affected / at risk) | 16/20 | 20/21
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/21
Other Adverse Events (participants affected / at risk) | 17/20 | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galinpepimut-S (N=20) | Control (N=21)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galinpepimut-S (N=20) | Control (N=21)
Injection site reaction (Surgical and medical procedures) | 17 (17) | 9 (9)
Fatigue (General disorders) | 10 (10) | 10 (10)
Fever (Immune system disorders) | 0 (0) | 4 (4)
Arthralgias (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Nausea (General disorders) | 2 (2) | 0 (0)
Rash, maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-07-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT01265433/Prot_SAP_ICF_000.pdf